CLINICAL TRIAL: NCT01555710
Title: A Multi-center, Open-Label, Adaptive, Randomized Study of Palifosfamide-tris, a Novel DNA Crosslinker, in Combination With Carboplatin and Etoposide (PaCE) Chemotherapy Versus Carboplatin and Etoposide (CE) Alone in Chemotherapy Naïve Patients With Extensive-Stage Small Cell Lung Cancer. The MATISSE Study
Brief Title: Study of Palifosfamide-tris in Combination With Carboplatin and Etoposide in Chemotherapy Naïve Patients With Extensive-Stage Small Cell Lung Cancer (The MATISSE Study)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPM3002
Record Dates: First submitted 2012-03-12; First posted 2012-03-15 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Extensive-Stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; isophosphamide mustard; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palifosfamide-tris plus Carboplatin and Etoposide (Experimental): Drug: palifosfamide-tris in combination with carboplatin and etoposide palifosfamide-tris: 130 mg/m2/day 3 days every 21 days for a max of 6 cycles. carboplatin: AUC 4 mg/mL/min 1 day every 21 days for a max of 6 cycles. etoposide: 100 mg/m2/day 3 days every 21 days for a max of 6 cycles.
  Interventions: Drug: Carboplatin; Drug: Palifosfamide-tris; Drug: Etoposide
- Carboplatin plus Etoposide (Active Comparator): Drug: carboplatin in combination with etoposide carboplatin: AUC 5mg/mL/min 1 day every 21 days for a maximum of 6 cycles. etoposide: 100 mg/m2/day 3 days every 21 days for a maximum of 6 cycles.
  Interventions: Drug: Etoposide; Drug: Carboplatin

INTERVENTIONS:
Drug: Carboplatin — AUC 4 mg/mL/min 1 day every 21 days for a max of 6 cycles.
  Arms: Palifosfamide-tris plus Carboplatin and Etoposide
Drug: Palifosfamide-tris — 130 mg/m2/day 3 days every 21 days for a max of 6 cycles.
  Arms: Palifosfamide-tris plus Carboplatin and Etoposide
Drug: Etoposide — 100 mg/m2/day 3 days every 21 days for a maximum of 6 cycles.
Drug: Carboplatin — AUC 5 mg/mL/min 1 day every 21 days for a max of 6 cycles.
  Arms: Carboplatin plus Etoposide

SUMMARY:
This is a multinational, multicenter, randomized controlled, open-label, adaptive study to evaluate the efficacy of PaCE chemotherapy in chemotherapy naive subjects with extensive-stage SCLC. Eligible subjects will be stratified according to age, gender, and Eastern Cooperative Oncology Group (ECOG) performance status, and randomized in a 1:1 ratio to receive either PaCE or CE chemotherapy.

The study design uses an adaptive group sequential approach with sample size re-estimation at the interim analysis.

Secondary efficacy endpoints include ORR, PFS, duration of response and changes in QOL and disease-related symptoms. Tumor-related endpoints will be assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guidelines.

The safety of study treatments will be assessed by the frequency and severity of adverse events as determined by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03. To provide an initial confirmation of safety, an early interim analysis of safety data only will be performed.

An independent Data Monitoring Committee (DMC) will be convened to assess the safety and efficacy of the study interventions and to monitor the overall conduct of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Documented extensive-stage small cell lung cancer.
* Patient has received no prior chemotherapy, adjuvant therapy, or radiotherapy for lung cancer.
* ECOG Performance Status of 0, 1 or 2.
* Adequate bone marrow and organ function based on the results of protocol- specified laboratory tests.
* Male and female patients must agree to use a highly reliable method of birth control during study participation.
* Able to provide informed consent

Exclusion Criteria:

* Previously untreated (non-irradiated), symptomatic brain metastases.
* Known allergy to any of the study drugs or their excipients.
* Any unstable or clinically significant concurrent medical condition that would, in the opinion of the investigator, jeopardize the safety of a patient and/or their compliance with the protocol, based on screening tests, physical examination and medical history (as specifically defined in the clinical protocol).
* Any malignancy other than small cell lung cancer within the last 5 years prior to randomization, with the exception of cervical carcinoma in situ, nonmelanoma skin cancer, or superficial bladder tumors (Ta, Tis, or T1) that have been successfully and curatively treated with no evidence of recurrent or residual disease. (Exception: Subjects with a history of malignancy other than small cell lung cancer may be enrolled after consultation with the medical monitor provided the patient's prognosis is best defined by the extensive-stage small cell lung cancer).
* Currently pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Assessed every 12 weeks for survival until 1 year following completion of enrollment

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Assessed every 6 weeks for 22 weeks, then every 12 weeks until progressive disease, initiation of alternate anticancer therapy, or 1 year following the last patient enrolled (whichever is soonest)
Quality of Life (QOL) as assessed by EQ-5D-3L and QLQ-LC13 | Assessed every 3 weeks for 22 weeks, then every 12 weeks until 1 year following the last patient enrolled
Objective Response Rate (ORR) | Assessed every 6 weeks for 22 weeks, then every 12 weeks until a partial or complete response is confirmed
Response Duration | Time from the date of first objective response (partial or complete response), with subsequent confirmation, until the date of disease progression or the occurrence of death
Safety parameters (number of adverse events as well as number of findings from physical examinations, ECGs, vital signs, and clinical laboratory results)using NCI CTCAE v. 4.03 | 22 weeks

CONTACTS AND LOCATIONS:
Locations (79):
- United States (40):
  - Birmingham Hematology and Oncology Associates, LLC, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - Redwood Regional Oncology Group, Santa Rosa, California
  - Christiana Care Health Services, Newark, Delaware
  - Baptist Cancer Institute, Jacksonville, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Sant Lucie, Florida
  - Peachtree Hematology Oncology Consultants, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Medical and Surgical Specialists, LLC, Galesburg, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Central Indiana Cancer Centers, Fishers, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University, Indianapolis, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Indiana University Health Ball Memorial Hospital, Muncie, Indiana
  - University of Kansas Hospital, Overland Park, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Medical Oncology, LLC, Baton Rouge, Louisiana
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - Metro Health Cancer Center, Wyoming, Michigan
  - Saint Mary's Medical Center, Duluth, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Hematology Oncology Associates of Northern New Jersey, PA, Carol G. Simon Cancer Center, Morristown, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New York Oncology Hematology, PC, Albany, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Dayton Cancer Center, Medical Oncology Hematology Associates, Dayton, Ohio
  - Medical Oncology Associates Of Wyoming Valley, PC, Kingston, Pennsylvania
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - Texas Oncology-Medical City Dallas, Dallas, Texas
  - Texas Oncology- Baylor, Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Oncology Consultants, PA, Houston, Texas
  - Texas Oncology, PA, Wichita Falls, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Fairfax Northern Virginia Hematology-Oncology, PC, Fairfax, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Wisconsin Institutes for Medical Research, Madison, Wisconsin
- Southern Medical Day Oncology Care Centre, Wollongong, New South Wales, Australia
- Canada (3):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - R. S. McLaughlin Durham Regional Cancer Center at Lakeridge Health Oshawa, Oshawa, Ontario
  - Hôpital Laval, Sainte-Foy, Quebec
- France (8):
  - Centre Hospitalier Lyon Sud, Pierre Bénité, Auvergne-Rhône-Alpes
  - Centre François Baclesse, Caen, Basse-normandie
  - Centre Hospitalier Universitaire -Hôpital Morvan, Brest, Brittany Region
  - Centre Hospitalier Universitaire, Hopital Bretonneau, Tours, Centre-Val de Loire
  - Hôpital du Cluzeau, Limoges, Limousin, Lorraine
  - Institut de Cancérologie de l'Ouest - René Gauducheau, Saint-Herblain, Pays de la Loire Region
  - Hôpital Saint Joseph, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Paul Strauss, Strasbourg
- Hungary (2):
  - Debreceni Egyetem Orvos és Egészségtudományi Centrum, Debrecen, Hajdú-Bihar
  - Mátrai Gyógyintézet, Mátraháza, Heves County
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Organization, Ein Kerem, Jerusalem
  - Meir Hospital Sapir Medical Center, Kfar Saba
  - Western Gallilee Medical Center, Nahariya
  - Rabin Medical Center Beilinson Campus, Petah Tikva
- Italy (3):
  - Istituto Nazionale per la Ricerca sul Cancro, Genova, Genova
  - Presidio Ospedaliero S. Chiara, Trento, Trento
  - Azienda Ospedaliera Ospedale Niguarda Ca' Granda, Milan
- Poland (4):
  - Centrum Onkologii - Instytut im. M. Sklodowskiej-Curie w Warszawie, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Wojewódzkie Centrum Onkologii, Gdansk, Pomeranian Voivodeship
  - Specjalistyczny Szpital im. Alfreda Sokolowskiego, Szczecin, West Pomeranian Voivodeship
- Russia (11):
  - Republic Clinical Oncology Dispensary of the Ministry of Healthcare of Republic of Bashkortostan, Ufa, Bashkortostan Republic
  - Ivanovo Regional Oncology Centre, Ivanovo, Ivanovo Oblast
  - City Oncology Hospital # 62, Moscow Region, Moscow
  - State Institution of Healthcare "Arkhangelsk Regional Clinical Oncology Dispensary", Arkhangelsk, Primorskiy (Maritime) Kray
  - Republican Clinical Oncologic Dispensary of Ministry of health of Republic Tatarstan, Kazan', Tatarstan Republic
  - State Budget Institution of Healthcare "Chelyabinsk Regional Clinical Oncology Dispensary", Chelaybinsk
  - Cancer Research Center n.a. N.N. Blokhin, Moscow
  - GUZ of Nizhegorodskiy region, Nizhnij Novgorod City Oncology Dispensary, Nizhny Novgorod
  - State Educational Institution "S.M. Kirov Military Medical Academy of Ministry of Defense of Russia", Saint Petersburg
  - Saint-Petersburg State Medical University n. a. I. P. Pavlov, Saint Petersburg
  - State healthcare institution of Yaroslavl region "Regional Clinical Oncologic Hospital", Yaroslavl
- China Medical University Hospital, Taichung, Taiwan
- Wythenshawe Hospital, Manchester, England, United Kingdom